CLINICAL TRIAL: NCT04976114
Title: Reducing Preoperative Anxiety in Parents of Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Emilio Vargas Castrillón, Head of clinical pharmacoloy hospital clinico san carlos, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: preoperative anxiety
Record Dates: First submitted 2021-07-09; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: A randomised and blind clinical trial. The parents could be randomly assigned to the control group, and received the standard procedure, or to the experimental groups. Three experimental groups were possible regarding the various types of interventions: story book (IG1), video (IG2), or both instruments (IG3)
Who Masked: Investigator
Masking Description: As it is not possible for the participants to be blinded, they were asked not to mention to the assessment researchers (or other parents they could meet) what was the information they received, ensuring the researchers to remain blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Standard of care
- story book (Experimental): Parents read a book with the chid previous to surgery.
  Interventions: Procedure: Story book with information about surgery techniques
- video (Experimental): Parents watch a video with the chid previous to surgery.
  Interventions: Procedure: Video with information about surgery techniques
- both instrument (Experimental): Parents read a book and watch a video with the chid previous to surgery.
  Interventions: Procedure: Story book and Video with information about surgery techniques

INTERVENTIONS:
Procedure: Story book with information about surgery techniques — Presurgery use of Story book. The parents with the child read a book with information about surgery techniques the days before surgery.
  Arms: story book
Procedure: Video with information about surgery techniques — Presurgery use of video. The parents with the child watch a video with information about surgery techniques the days before surgery.
  Arms: video
Procedure: Story book and Video with information about surgery techniques — Presurgery use of video and story book. The parents with the child watch a video and read a book (both) with information about surgery techniques the days before surgery.
  Arms: both instrument

SUMMARY:
Aims and objectives: To investigate preoperative anxiety in parents of paediatric surgical patients, testing whether the provision of information (using video and story books) regarding the surgical process can impact on reducing anxiety. Analyse if some personal factors influence the reduction of anxiety.

Background: Attending a surgical theatre generates anxiety in all types of patients, especially in the case of children. The effect of different preoperative intervention procedures in children that attempt to reduce their anxiety level have been studied a great deal. However, although their parents also suffer high anxiety levels, potential intervention to reduce their levels have not received the same attention.

Study design: Randomised Clinical trial Methods: One hundred and twenty-five parents of children (8-12 y.o.) undergoing surgery in Hospital Universitario Central de Asturias hospital (Oviedo, Spain) were randomly assigned to the control group (34 individuals) or one of the 3 experimental groups (91). After the pre-anaesthesia consultation, children and parents of the experimental groups were provided with a story book, a video with additional information of nursing, or both. In the antechamber of the operating room and prior to the surgical intervention, the State Anxiety and Trait Anxiety of the parents and children were measured using the STAI and STAIC questionnaires respectively. The data collection, including different demographic variables was carried out for 12 months starting in October 2016

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery at Asturias Central Hospital

Exclusion Criteria:

* Children not in the age range,
* Emergency surgery,
* Children not able to understand or read
* Parents not present or refused to participate.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Anxiety level | Presurgery, just the moment before to surgery
  Level of presurgery anxiety measured by State-Trait Anxiety Inventory scale

IPD SHARING:
Plan to Share IPD: No
The results will be able after request with considerable reasons